CLINICAL TRIAL: NCT04215757
Title: PERIPHERAL NERVE BLOCKS WITH LOW DOSE LIGNOCAINE FOR THE TREATMENT OF ACUTE LUMBOSACRAL RADICULOPATHY
Brief Title: Low Dose Lignocaine Injections as a Treatment Option for Acute Lumbosacral Radiculopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences, Rishikesh (Other Government)
Responsible Party: Principal Investigator, ADABALA VIJAY BABU, Principal Investigator, All India Institute of Medical Sciences, Rishikesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patient received one or two peripheral nerve blocks at a maximum according to their involvement in the operation theatre, with full ASA monitoring under all aseptic precautions.
  For L4 radiculopathy Saphenous nerve block with 1.5ml of 2% lignocaine diluted to 10ml (0.3%) For L5 radiculopathy Deep peroneal nerve block/posterior tibial nerve block with 1.5ml of 2% lignocaine diluted to 10ml (0.3%) For S1 radiculopathy Sural nerve block with 1.5ml of 2% lignocaine diluted to 10ml (0.3%)
  Interventions: Procedure: peripheral nerve block
- Control group (Placebo Comparator): Patients received one or two peripheral nerve blocks at a maximum according to their involvement in the operation theatre, with full ASA monitoring under all aseptic precautions.
  For L4 radiculopathy Saphenous nerve block with 10ml distilled water For L5 radiculopathy Deep peroneal nerve block/posterior tibial nerve block with 10ml distilled water For S1 radiculopathy Sural nerve block with10ml distilled water
  Interventions: Procedure: peripheral nerve block

INTERVENTIONS:
Procedure: peripheral nerve block — peripheral nerve blocks with low dose lignocaine in acute radiculopathy

SUMMARY:
Low back pain is one of the most common ailments that plagues patients, with nearly 80% of the population developing some form of back pain in their lifetime. Up regulated sodium channels in the nerve root or dorsal root ganglion are the basic cause for the mechano-sensitization and injecting the drug in the peripheral end of the nerve will block these sodium channels, since functionally both ends of the pseudo unipolar neuron are the same.

DETAILED DESCRIPTION:
Low back pain is one of the most common ailments that plague patients, with nearly 80% of the population developing some form of back pain in their lifetime. Of all the causes of low back pain, the most common is lumbar radicular pain which may result from irritation of the nerve fibers or dorsal root ganglia due to intervertebral disc prolapse, degenerative spondylolisthesis or spinal canal stenosis. [1] Up regulated sodium channels in the nerve root or dorsal root ganglion are the basic cause for the mechano-sensitization and injecting the drug in the peripheral end of the nerve will block these sodium channels, since functionally both ends of the pseudo unipolar neuron are the same. [2]There have yet been no studies done to prove the efficacy of peripheral nerve block as an alternative to lumbar epidurals. We would like to share our experience of peripheral nerve blocks with low dose local Anaesthetics as the treatment of acute lumbosacral radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 years to 60 years
* Pain involving up to two segmental levels (L4, L5 and S1).
* Average pain score of ≥5 on an 11-point NRS.
* Tenderness over the concordant peripheral nerves (Gore sign +)
* Computed tomography/Magnetic resonance imaging evidence of nerve root pain concordant with the side and level of clinical features.

Exclusion Criteria:

* Coagulopathy and/or patients on anticoagulants.
* Infection at the site of injection.
* Hypersensitivity to a local anaesthetic agent.
* Evidence of significant sensory or progressive motor deficit.
* Presence of cancer as a cause of back pain.
* History of previous backs surgery/epidural steroid injection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-20 (Actual); Primary Completion 2020-01-15 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
≥50% or ≥4 point reduction in an 10-point numeric scale (NRS) at, 1 month, 2 months and 3 months. | 3 months
  change in pain intensity measured with numeric scale.Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an ten-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Adabala, MD, Principal Investigator — AIIMS Rishikesh
Locations (1):
- AIIMS, Rishikesh, Uttarakhand, India

IPD SHARING:
Plan to Share IPD: Yes
once the study is finished
Supporting Information: Study Protocol, CSR
Time Frame: 6 months
Access Criteria: on web

REFERENCES:
- [Result] Levinson SR, Luo S, Henry MA. The role of sodium channels in chronic pain. Muscle Nerve. 2012 Aug;46(2):155-65. doi: 10.1002/mus.23314. PMID 22806363